CLINICAL TRIAL: NCT00336713
Title: A Multicenter, 24-52-week, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, and Safety of Saredutant 100 mg Once Daily in the Prevention of Relapse of Depressive Symptoms in Outpatients With Major Depressive Disorder
Brief Title: A 24-52-week Study to Evaluate the Long-term Efficacy and Safety of Saredutant in Patients With Depression (MAGENTA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5576; SR48968
Record Dates: First submitted 2006-06-13; First posted 2006-06-14 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-04

CONDITIONS: Depressive Disorder
Keywords: depression; antidepressive agents; controlled clinical trial
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — SR 48968

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saredutant 100 mg (Experimental): Saredutant 100 mg once daily in the morning for a maximum of 64 weeks
  Interventions: Drug: Saredutant (SR48968C)
- Placebo (Placebo Comparator): Placebo for Saredutant once daily in the morning during the maintenance phase for a maximum of 52 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saredutant (SR48968C) — oral administration (capsules)
  Arms: Saredutant 100 mg
Drug: Placebo — oral administration (capsules)
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the long-term efficacy and safety of Saredutant in patients with depression. The primary objective is to evaluate the efficacy and safety of Saredutant 100 mg once daily compared to placebo in the prevention of relapse of depressive symptoms in outpatients with major depressive disorder who achieved an initial response to 12 weeks of open-label treatment with Saredutant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder, as defined by Diagnostic and Statistical Manual of Mental Disorders 4th edition (DSM-IV) criteria and confirmed by the semi-structured Mini International Neuropsychiatric Interview (MINI), recurrent episode.

Exclusion Criteria:

* Total score of 28 or less on the Montgomery and Asberg Depression Rating Scale (MADRS).
* Clinical Global Impression (CGI) severity score of less than 4.
* Duration of the current depressive episode less than 2 months or greater than 2 years.
* Elderly patients with a Mini-Mental State Examination (MMSE) total score <25.
* Patients with a history or presence of bipolar disorders or psychotic disorders.
* Patients with alcohol dependence or abuse or substance dependence or abuse in the past 12 months except nicotine or caffeine dependence.
* Benzodiazepine or sedative-hypnotic use greater than 2 days per week during the month prior to entry into the Acute Phase.
* Patients who have used the following prior to entry into Acute Phase: antipsychotics within 3 months, fluoxetine within 1 month, Monoamine oxidase inhibitors (MAOIs) within 2 weeks, other antidepressant or mood-stabilizer (lithium, anticonvulsants) within 1 week.

The investigator will evaluate whether there are other reasons why a patient may not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2006-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The time to relapse of depressive symptoms (in days) during the Maintenance Phase. | minimum 24 weeks and maximum 52 weeks

SECONDARY OUTCOMES:
Changes from baseline in the CGI Severity of Illness, Montgomery-Asberg Depression Rating Scale (MADRS) total, and Hamilton Anxiety Rating Scale (HAM-A) total and factor scores during the Maintenance Phase. | minimum 24 weeks and maximum 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States